CLINICAL TRIAL: NCT01025544
Title: A Phase III Open Label, Multi-Center Pediatric Study in China Comparing Booster Doses of Vaxem Hib and Hiberix Vaccines for the Prevention of Haemophilus Influenzae Type b (Hib) Infection
Brief Title: Study in Toddlers (12-18 Months) Comparing a Booster Dose of Vaxem Hib and Hiberix Vaccines for the Prevention of Haemophilus Influenzae Type b Infections in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M37P2E1
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Haemophilus Influenzae Type b (Hib) Infection
Keywords: Haemophilus influenzae type b (Hib); Vaccine; Booster
MeSH Terms: conditions — Haemophilus Infections; Infections | interventions — Vaccines; Hiberix

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Biological: Vaxem Hib (Haemophilus influenzae type b (Hib) vaccine)
- Arm 2 (Active Comparator)
  Interventions: Biological: Hiberix (Haemophilus influenzae type b (Hib) vaccine)

INTERVENTIONS:
Biological: Vaxem Hib (Haemophilus influenzae type b (Hib) vaccine) — Comparator study of two commercially available Haemophilus influenzae type b (Hib) vaccines.
  Arms: Arm 1
Biological: Hiberix (Haemophilus influenzae type b (Hib) vaccine) — Comparator study of two commercially available Haemophilus influenzae type b (Hib) vaccines.
  Arms: Arm 2

SUMMARY:
This study will evaluate the safety and immunogenicity of booster doses of the two vaccines used to prevent Haemophilus influenzae type b infections in children 12-18 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Toddlers 12-18 months of age who have previously participated in study M37P2.

Exclusion Criteria:

* Prior Hib booster administration.
* History of serious reaction(s) following vaccination.
* Vaccination within 14 days of study vaccination.
* Known or suspected immune impairment.
* For additional entry criteria please refer to the protocol.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 846 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Anti-PRP antibody levels at day 31 post booster | 31 days after vaccination

SECONDARY OUTCOMES:
Solicited local and systemic reactions, AEs, and SAEs | 30 days post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Basel, Study Chair — 41 61 324 1111
Locations (1):
- Hebei Province, China